CLINICAL TRIAL: NCT06894043
Title: Effect of an Intervention Program of Adapted Physical Activity Combined With Compensatory Nutrition in Patients With Constitutional Thinness
Acronym: ANIMATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire Interuniversitaire de Biologie de la Motricité (Other); Target Tape (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24CH263; ANSM (Other: 2025-A00088-41)
Record Dates: First submitted 2025-02-04; First posted 2025-03-25 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Constitutional Thinness
Keywords: Constitutional thinness (CT); Adapted Physical Activity; Compensatory nutrition; Lean and muscle mass gain; Resistance to gain weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APA + NC (Experimental)
  Interventions: Other: Adapted Physical Activity (APA); Behavioral: Compensatory Nutrition (NC)
- Control (No Intervention): * 2-week run-in period
  * Followed by an 8-week period of conventional management without APA and without NC

INTERVENTIONS:
Other: Adapted Physical Activity (APA) — The APA intervention will consist of a 2-week running-in period, followed by a period of adapted physical activity (APA) for 8 weeks.
  Arms: APA + NC
Behavioral: Compensatory Nutrition (NC) — The Compensatory Nutrition (NC) intervention will consist of a 2-week running-in period, followed by a period of compensated nutrition (NC) for 8 weeks.
  Arms: APA + NC

SUMMARY:
Constitutional Thinness (CT) is a form of stable thinness without malnutrition but with resistance to weight gain, affecting approximately 1% of the general population. The clinical consequences are numerous and the pathophysiology remains poorly understood.

Currently, conventional management involves a high-calorie and frequent diet, combined with the avoidance of endurance physical activity, although there is no significant evidence of its effectiveness.

Our hypothesis is that an adapted physical activity program (APA) combined with compensatory nutrition (CN) could help these patients gain lean mass (muscle mass).

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female
* BMI: ≤ 18.5 kg/m²
* Weight Stability: Stable weight for at least 3 months
* Age: 18 to 50 years old at the inclusion visit
* Diagnosed with Constitutional thinness

Exclusion Criteria:

* Pregnancy, Parturition, or Lactation
* Legal Restrictions: Individuals deprived of liberty, involuntarily hospitalized, or hospitalized for reasons other than research purposes, adults under legal protection (guardianship or curatorship) or unable to provide consent
* Eating Disorders: Individuals with eating disorders (DSM IV and 5 criteria)
* Excessive Alcohol Consumption: Consumption exceeding the equivalent of 10 glasses of wine per week
* Severe Progressive Conditions: Progressive severe conditions (e.g., diabetes)
* Intense Physical Activity: Individuals engaging in intense physical activity (> 3 sessions per week)
* Heavy Smoking: Significant smoking (>10 cigarettes per day)
* Psychiatric Conditions: Presence of depressive or psychiatric conditions requiring antidepressant or psychotropic treatment
* Medical or Surgical History: Medical or surgical history deemed incompatible with the study by the investigator
* MRI Contraindication: Individuals with contraindications to MRI will not undergo spectro-MRI analyses

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Lean body mass | From day 1 to week 8
  Lean body mass gain (kg) measured by bioimpedance

SECONDARY OUTCOMES:
BMI | From day 1 to week 8
  Body masse index : ratio between weight and height
Energy balance | From day 1 to week 8
  Ratio between calorie intake and calorie expenditure
  Caloric intake measured by dietary records over 2 weeks (calorie); Calorie expenditure: Resting metabolism measured by indirect calorimetry (kcal/24h); + Postprandial thermogenesis measured by indirect calorimetry (kcal/24h);; + Physical activity energy expenditure measured by connected watch (kcal/24h);
Physical exercise capacity | From day 1 to week 8
  Changes in VO2max
Quality of life SF-12 questionnaire | From day 1 to week 8
  SF-12 questionnaire; Self-measurement questionnaire SF-12 (Short Form Health Survey 12); comprising 12 questions assessing 8 dimensions, namely physical functioning, role limitation due to physical problems, role limitation resulting from emotional problems, vitality (energy/fatigue), emotional well-being, social functioning, bodily pain, and perception of general and mental health; each dimension is represented by a score ranging from 0 to 100, with a low score signifying poor health perception in the dimension considered, and a high score signifying the opposite);

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France, France